CLINICAL TRIAL: NCT05235152
Title: Group-based Exercise Training Programs for Military Members Presenting Musculoskeletal Disorders - A Pragmatic Randomized Controlled Trial
Brief Title: Group-based Exercise Training Programs for Military Members With Musculoskeletal Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-2039
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Musculoskeletal Pain; Low Back Pain; Rotator Cuff Tendinitis; Patellofemoral Pain Syndrome; Ankle Sprains
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain; Rotator Cuff Injuries; Patellofemoral Pain Syndrome; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized-controlled trial with four evaluation sessions over 26 weeks (baseline, week 6 [mid-intervention], week 12 [end of intervention], week 26) and 16 visits over 12 weeks to the Valcartier Health Centre for the intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research assistant and treating therapist will be blinded to baseline evaluation results. Given that for this type of intervention it is impossible to blind the treating physiotherapists and participants, only the investigator, evaluator and statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual individual physiotherapy care (Active Comparator): Participants with either low back pain, rotator cuff related pain, patellofemoral pain syndrome or lateral ankle sprain will received usual/individual physiotherapy care over a period of 12-weeks for the treatment of their musculoskeletal conditions if randomized in this group.
  Interventions: Other: Usual individual physiotherapy care
- Group-supervised physiotherapy training programs (Experimental): Participants with either low back pain, rotator cuff related pain, patellofemoral pain syndrome or lateral ankle sprain will received group-supervised physiotherapy training programs over a period of 12-weeks for the treatment of their musculoskeletal condition if randomized in this group.
  Interventions: Other: Group-supervised physiotherapy training programs

INTERVENTIONS:
Other: Usual individual physiotherapy care — Usual and individual physiotherapy care guidelines were developed through a round-table discussion involving experts in musculoskeletal health. From the round-table discussion, the consensus as reflecting best-practices for the rehabilitation of musculoskeletal rehabilitation supported an active exercise rehabilitation approach which includes strengthening and neuromuscular training exercises. Furthermore, the following treatments are considered in addition to active exercises:
  * Range of motion: active, active-assisted, passive, repeated movements (Mulligan or McKenzie);
  * Stretching / manual therapy: mobilizations, manipulation, neural mobility, active release therapy;
  * Individual proprioceptive training.
  Arms: Usual individual physiotherapy care
Other: Group-supervised physiotherapy training programs — Three group-supervised physiotherapy training programs (The lumbar, the upper extremity and the lower extremity training programs) were developed for military members with musculoskeletal conditions. They are composed of stations that each include several exercises of varying levels of difficulty. Group size will vary between 5 to 20 participants for one physiotherapist, and each military member performs his/her own exercises. During a typical session, the participant and therapist will choose one exercise to perform per station according to two main criteria: severity of the condition and the ability to perform the exercises optimally. The level of supervision is adapted to the participant's needs and performance. Progression in the programs leads to the execution of exercises that simulate functional and occupational tasks.
  Arms: Group-supervised physiotherapy training programs

SUMMARY:
This randomized controlled trial will compare the mid- and long-term effects of group-based training programs with usual individual physiotherapy care for the treatment of musculoskeletal disorders in military. One hundred and twenty soldiers presenting one of the four targeted musculoskeletal disorders (low back pain, rotator cuff related pain, patellofemoral pain syndrome or lateral ankle sprain) will be recruited and randomly assigned to either a 12-weeks group-based training program or 12-weeks usual individual physiotherapy care.

DETAILED DESCRIPTION:
Musculoskeletal disorders are a leading cause of morbidity and the most prevalent source of disability among soldiers. Their high prevalence in armed forces and limited resources have led to problems related to access to physical rehabilitation care. To increase access, supervised group-based exercise programs for the most prevalent musculoskeletal disorders (low back pain, patellofemoral pain, rotator cuff-related shoulder pain or lateral ankle sprain) have been developed at a Canadian Armed forces (CAF) base, but their effectiveness has not been evaluated. The primary objective of this randomized controlled trial is to evaluate the mid- and long-term effects of these group-based training programs on pain severity and functional limitations, in comparison with usual individual physiotherapy care. Secondary objectives include comparing both interventions in terms of health-related quality of life, pain-related fear, and patients' satisfaction.

One hundred and twenty soldiers with a new medical referral for physiotherapy services for one of the four targeted musculoskeletal disorders will be consecutively recruited. They will be randomly assigned to either group-based training program or usual individual physiotherapy care, and will take part in the assigned 12-week intervention. There will be four evaluation sessions over 26 weeks (baseline, week 6, 12 and 26). At each follow-up, functional limitations, pain severity, health-related quality of life and pain-related fears will be assessed. Patients satisfaction with treatment will also be evaluated at the end of the intervention period. A two-way repeated measures ANOVA will be used to analyze and compare the effects of the interventions.

The results of this randomized controlled trial will determine the effectiveness of group-based training programs compared to usual individual physiotherapy care. This new intervention model could represent an efficient, and more pro-active approach to manage a higher number of soldiers with musculoskeletal disorders. It could improve access to physical rehabilitation care and improve the health of soldiers.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-60 years
* Present one of the four targeted musculoskeletal disorders:

Low back pain:

Inclusion - 1) Low back pain with or without radiation to the lower limbs, 2) minimal score of 17% on the Modified Oswestry Disability Index (ODI).

Exclusion - 1) history of surgery or fracture to the spinal column, 2) signs of upper motor neuron lesions (bilateral paresthesia, hyperreflexia or spasticity) or other red flags (e.g. fracture).

Patellofemoral pain syndrome:

Inclusion - 1) anterior knee pain during running or during at least two activities among: kneeling, squatting, and resisted knee extension 2) score lower than 85/100 on the Knee Outcomes Survey - Activity of Daily Living Scale (KOS- ADLS).

Exclusion - 1) history of knee surgery or patellar dislocation; 2) pain believed to originate either from meniscus (presence of joint line fullness and tenderness, McMurray sign, and positive Thessaly test) or from any knee ligament.

Rotator cuff-related shoulder pain:

Inclusion - 1) at least one positive finding in each of the following categories: a) painful arc of movement; b) positive Neer's or Kennedy-Hawkins Test; c) pain on resisted external rotation, resisted abduction or Empty Can Test 2) minimal score of 14 points on the Disabilities of the Arm, Shoulder and Hand (QuickDASH).

Exclusion - 1) history of shoulder surgery, fracture, capsulitis, or dislocation, 2) full thickness rotator cuff tear identified by imagery or clinical tests 3) cervicobrachialgia or shoulder pain reproduced by neck movements.

Lateral ankle sprain:

Inclusion - 1) unilateral lateral ankle sprain of <6 weeks, 2) minimal score of 9 points on the Lower Extremity Functional Scale (LEFS).

Exclusion - 1) ankle fracture, 2) lateral ligaments not the principal injury (a high ankle/tibiofibular sprain).

Exclusion Criteria for all diagnosis:

1. Are unavailable to participate in a 12-week intervention;
2. Have a diagnosis of rheumatoid, inflammatory, neurological or neurodegenerative disease;
3. Received a corticosteroid injection in the previous 6 weeks in the affected region;
4. Have had more than 6 months of work restriction for their current musculoskeletal pain;
5. Acute conditions (Constant and intense pain [>5/10];Severely limited range of motion [more than 50% in at least 2 directions]; Obvious lateral shift for low back pain or Unable to bear weight [for lateral ankle sprain])

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional limitations | Week 26
  Pain-related functional limitations will be measured with the Pain Interference subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Interference subscale is recommended for assessment of pain-related functional limitations and includes seven items that measure the level of interference with function caused by pain using 0 (no interference) to 10 (complete interference) rating scales.

SECONDARY OUTCOMES:
Functional limitations | Week 6 (mid-intervention)
  Pain-related functional limitations will be measured with the Pain Interference subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Interference subscale is recommended for assessment of pain-related functional limitations and includes seven items that measure the level of interference with function caused by pain using 0 (no interference) to 10 (complete interference) rating scales.
Functional limitations | Week 12 (end of intervention)
  Pain-related functional limitations will be measured with the Pain Interference subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Interference subscale is recommended for assessment of pain-related functional limitations and includes seven items that measure the level of interference with function caused by pain using 0 (no interference) to 10 (complete interference) rating scales.
Pain severity | Week 6 (mid-intervention)
  Pain severity will be measured with the Pain Severity subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Severity subscale of the BPI includes four items that measure pain intensity using 0 (no pain) to 10 (pain as bad as you can imagine) rating scales.
Pain severity | Week 12 (end of intervention)
  Pain severity will be measured with the Pain Severity subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Severity subscale of the BPI includes four items that measure pain intensity using 0 (no pain) to 10 (pain as bad as you can imagine) rating scales.
Pain severity | Week 26
  Pain severity will be measured with the Pain Severity subscale of the Brief Pain Inventory - Short Form (BPI). The Pain Severity subscale of the BPI includes four items that measure pain intensity using 0 (no pain) to 10 (pain as bad as you can imagine) rating scales.
Health-related quality of life | Week 6 (mid-intervention)
  Health-related quality of life will be measured with the five-level version of EQ-5D (EQ-5D-5L). The EQ-5D-5L is a generic health-related quality of life (HRQoL) questionnaire that contains five questions covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question is rated on a five-point scale from 1 (no problems) to 5 (unable to perform). The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score ranging from 0 to 1.
Health-related quality of life | Week 12 (end of intervention)
  Health-related quality of life will be measured with the five-level version of EQ-5D (EQ-5D-5L). The EQ-5D-5L is a generic health-related quality of life (HRQoL) questionnaire that contains five questions covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question is rated on a five-point scale from 1 (no problems) to 5 (unable to perform). The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score ranging from 0 to 1.
Health-related quality of life | Week 26
  Health-related quality of life will be measured with the five-level version of EQ-5D (EQ-5D-5L). The EQ-5D-5L is a generic health-related quality of life (HRQoL) questionnaire that contains five questions covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question is rated on a five-point scale from 1 (no problems) to 5 (unable to perform). The combined dimensions describe 55 = 3125 theoretically possible states of health that can be converted into a weighted index score ranging from 0 to 1.
Pain-related fear | Week 6 (mid-intervention)
  Pain-related fear will be measured with the Tampa scale of kinesiophobia. The Tampa scale of kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided.
Pain-related fear | Week 12 (end of intervention)
  Pain-related fear will be measured with the Tampa scale of kinesiophobia. The Tampa scale of kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided.
Pain-related fear | Week 26
  Pain-related fear will be measured with the Tampa scale of kinesiophobia. The Tampa scale of kinesiophobia is a 11-item scale measuring beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided.
Satisfaction with treatment - PASS | Week 12 (end of intervention)
  Patients satisfaction with treatment will be assessed using the Patient Acceptable Symptom State (PASS). It asks patients if they are satisfied with their current state or not and to rate their satisfaction on a 0-10 numeric scale (0 representing not satisfied at all, and 10 very much satisfied).
Satisfaction with treatment - Likert Scale | Week 12 (end of intervention)
  Participants will be asked to rate their satisfaction with treatment received using a three-item Likert scale (''not satisfied'', ''satisfied'' or ''very much satisfied''), their satisfaction with the frequence of treatments (''not enough'', ''just right'' or ''too much''), their satisfaction with the duration of treatments (''too short'', ''long enough''or ''too long'') and their satisfaction with the time spent with the physical therapist during the treatments ("not enough'', ''just right'' or ''too much'').
Low back pain-specific symptoms and functional limitations | Week 6
  Low back pain-specific symptoms and functional limitations will be evaluated for soldiers with low back pain with the Oswestry Disability Index (ODI) questionnaire. The ODI is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living using 0 (no difficulty) to 5 (incapacity) rating scales.
Low back pain-specific symptoms and functional limitations | Week 12
  Low back pain-specific symptoms and functional limitations will be evaluated for soldiers with low back pain with the Oswestry Disability Index (ODI) questionnaire. The ODI is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living using 0 (no difficulty) to 5 (incapacity) rating scales.
Low back pain-specific symptoms and functional limitations | Week 26
  Low back pain-specific symptoms and functional limitations will be evaluated for soldiers with low back pain with the Oswestry Disability Index (ODI) questionnaire. The ODI is a 10-item questionnaire that assesses the interference of low back pain with activities of daily living using 0 (no difficulty) to 5 (incapacity) rating scales.
Shoulder disorders-specific symptoms and functional limitations | Week 6
  Shoulder-specific symptoms and functional limitations will be evaluated for soldiers with rotator cuff related pain using the shortened version of the Disabilities of the Arm, Shoulder and Hand (QuickDASH). It is an 11-item questionnaire addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs using 0 (no difficulty or no symptoms) to 5 (incapacity or important symptoms) rating scales.
Shoulder disorders-specific symptoms and functional limitations | Week 12
  Shoulder-specific symptoms and functional limitations will be evaluated for soldiers with rotator cuff related pain with the shortened version of the Disabilities of the Arm, Shoulder and Hand (QuickDASH). It is an 11-item questionnaire addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs using 0 (no difficulty or no symptoms) to 5 (incapacity or important symptoms) rating scales.
Shoulder disorders-specific symptoms and functional limitations | Week 26
  Shoulder-specific symptoms and functional limitations will be evaluated for soldiers with rotator cuff related pain with the shortened version of the Disabilities of the Arm, Shoulder and Hand (QuickDASH). It is an 11-item questionnaire addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs using 0 (no difficulty or no symptoms) to 5 (incapacity or important symptoms) rating scales.
Knee disorders-specific symptoms and functional limitations | Week 6
  Knee-specific symptoms and functional limitations will be evaluated for soldiers with patellofemoral pain syndrome using the Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS). It is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations experienced during activities of daily living in individuals with various knee disorders using 5 (no difficulty) to 0 (incapacity) rating scales.
Knee disorders-specific symptoms and functional limitations | Week 12
  Knee-specific symptoms and functional limitations will be evaluated for soldiers with patellofemoral pain syndrome using the Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS). It is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations experienced during activities of daily living in individuals with various knee disorders using 5 (no difficulty) to 0 (incapacity) rating scales.
Knee disorders-specific symptoms and functional limitations | Week 26
  Knee-specific symptoms and functional limitations will be evaluated for soldiers with patellofemoral pain syndrome using the Knee Outcome Survey Activities of Daily Living Scale (KOS-ADLS). It is a 14-item knee-specific questionnaire that evaluates symptoms and functional limitations experienced during activities of daily living in individuals with various knee disorders using 5 (no difficulty) to 0 (incapacity) rating scales.
Ankle disorders-specific symptoms and functional limitations | Week 6
  Ankle-specific symptoms and functional limitations will be evaluated for soldiers with lateral ankle sprain using the Lower Extremity Functional Scale (LEFS). It is a 20-item questionnaire assessing the impairment of the lower-extremity musculoskeletal system in everyday activities using a 0 (incapacity) to 4 (no difficulty) rating scale.
Ankle disorders-specific symptoms and functional limitations | Week 12
  Ankle-specific symptoms and functional limitations will be evaluated for soldiers with lateral ankle sprain using the Lower Extremity Functional Scale (LEFS). It is a 20-item questionnaire assessing the impairment of the lower-extremity musculoskeletal system in everyday activities using a 0 (incapacity) to 4 (no difficulty) rating scale.
Ankle disorders-specific symptoms and functional limitations | Week 26
  Ankle-specific symptoms and functional limitations will be evaluated for soldiers with lateral ankle sprain using the Lower Extremity Functional Scale (LEFS). It is a 20-item questionnaire assessing the impairment of the lower-extremity musculoskeletal system in everyday activities using a 0 (incapacity) to 4 (no difficulty) rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University, Quebec, Qc (Canada)
Locations (1):
- Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupuis F, Perreault K, Hebert LJ, Perron M, Fredette MA, Desmeules F, Roy JS. Group-based exercice training programs for military members presenting musculoskeletal disorders - protocol for a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2022 Apr 18;23(1):366. doi: 10.1186/s12891-022-05317-6. PMID 35436907